CLINICAL TRIAL: NCT02788994
Title: Outcome Following Stabilization of Fresh Unilateral Unstable Pertrochanteric Hip Fracture With Either the Endovis BA2 Cephalomedullary Nail or the Dynamic Hip Screw: A Single Centre, Feasibility Study
Brief Title: Stabilization of Fresh Unilateral Unstable Pertrochanteric Hip Fracture
Acronym: PET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: Citieffe S.r.l (Industry)
Responsible Party: Principal Investigator, PeterGiannoudis, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OR15/280
Record Dates: First submitted 2015-09-11; First posted 2016-06-02 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Unilateral Unstable Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endovis BA2 Nail (Experimental): The EBA2 intramedullary nailing system is designed for the treatment of lateral proximal femoral fractures, and consists of a standard or medium length nail implantable with the same set of instruments.
  The system has been designed to allow:
  * stable fracture synthesis for fast rehabilitation and early mobilization
  * an efficient set of instruments (only 11) for a swift, reproducible operating technique (just 7 surgical steps)
  This is a one off surgical fixation.
  Interventions: Device: Endovis BA2 nail
- Dynamic Hip Screw (DHS) (Active Comparator): The DHS is designed to provide strong and stable internal fixation of a variety of intertrochanteric, subtrochanteric and basilar neck fractures, with minimal soft tissue irritation.
  This Dynamic Hip Screw method is currently used and is a one off surgical fixation.
  Interventions: Device: Dynamic Hip Screw (DHS)

INTERVENTIONS:
Device: Endovis BA2 nail — The EBA2 intramedullary nailing system is designed for the treatment of lateral proximal femoral fractures, and consists of a standard or medium length nail implantable with the same set of instruments.
  The system has been designed to allow:
  * stable fracture synthesis for fast rehabilitation and early mobilization
  * an efficient set of instruments (only 11) for a swift, reproducible operating technique (just 7 surgical steps)
  Arms: Endovis BA2 Nail
Device: Dynamic Hip Screw (DHS) — The DHS is designed to provide strong and stable internal fixation of a variety of intertrochanteric, subtrochanteric and basilar neck fractures, with minimal soft tissue irritation.
  This Dynamic Hip Screw method is currently used and is a one off surgical fixation.
  Arms: Dynamic Hip Screw (DHS)

SUMMARY:
This is a preliminary study to establish the issues and potential of the investigators proposed project, which involves recruitment of patients with and without dementia, who have been admitted to hospital following hip fractures. The study will be evaluating the result of treatment of unstable pertrochanteric hip fractures focusing on how soon mobility is restored leading to their independence. These patients would require surgical fixation (not replacement) of their hip fractures.

The study will evaluate two methods of fixation of hip fractures treated with either a pin (nail) which is inserted within the cavity of the thigh bone or a hip screw with a plate which is applied on the outer aspect of the thigh bone.

The data collected from this study will provide information on whether one method of fixation is better than the other.

DETAILED DESCRIPTION:
The investigators have organised a Patient Feedback Session in Leeds, comprising of patients who previously sustained hip fractures and who underwent surgical fixation (either cephalomedullary nail or dynamic/sliding hip screw). According to the feedback that was provided, the most important issue highlighted was how quickly the patients regain their functional capacity (mobility) and by inference their independence and overall quality of life, to pre-injury levels. The length of hospital stay was also an important parameter in their judgement.

Based on this patient feedback session, the design of a study evaluating the result of treatment of unstable pertrochanteric hip fractures should focus on how soon mobility is restored leading to their independence. Moreover, using the length of hospital stay as a secondary outcome would not only act as a surrogate of mobility (hospital discharge is determined by ability to safely mobilize), but would have huge implication to health care cost as well, which is considered as a major contributor for the majority of the overall hospital costs. Finally, it has been shown that up to 50% of hip fracture patients have dementia, which has been reported to be an independent risk factor of poor outcome following hip fractures. The investigators can therefore argue that it is even more important that this cohort of patients be treated with a superior implant, and thus be included in studies. However, currently, there is limited experience with regards to clinical trials which involve surgical patients with dementia, particularly on issues of consent, recruitment and retention/follow-up. This was highlighted by a recent review, who found that 8 out of 10 hip fracture trials excluded or ignored the patient population with cognitive impairment. However, with up to one in three patients with hip fractures presenting simultaneously with some degree of dementia, this is an important population to include.

The investigators therefore propose concept feasibility study, to investigate the feasibility of running a study involving patients with and without dementia to investigate the outcome of unstable pertrochanteric fractures (AO/OTA type A2), comparing the implantation of the Endovis BA 2 cephalomedullary nail (device conferring biomechanical advantage) to the Dynamic/Sliding Hip Screw (current "gold standard").

Patients who fulfill the inclusion and exclusion criteria, will be invited to participate in this study. Following patient or patient's carer/personal or nominated consultee providing informed consent/assent to participate in the study they will be randomized using an online randomisation tool, by permuted blocks, stratified for cognitive status (AMTS<8/≥8).

The abbreviated mental test score (AMTS) can rapidly assess elderly patients for the possibility of dementia and can assess for confusion and other cognitive impairment. The doctor seeing the patient will conduct the AMTS as standard of care.

Although patients will not be told of their allocation but cannot be considered blinded as they may guess which group they have been allocated based on the incision size. The assessor for clinical outcomes, such as the TUG assessment will be blinded to group allocation.

Following surgery, patients will be followed-up at week 2, 4 and 12 post-operation (as per standard of care practice). Information collected during these visits will include, hip X-rays, functional scores (Lower Extremity Measure, London Handicap Scale, DEMQOL), TUG (Timed Up and Go) test, complications/adverse events and concomitant medication requirements.

Within standard care patients undergo the above stages, the only extra measures with this research project from the above are the Lower Extremity measure, London Handicap Scale and TUG test.

Lower Extremity Measure will be used on patients with AMTS score ≥8 only whereas London Handicap Scale will be used on patients with AMTS score ≥8 only.

The TUG test involves standing up from a seated position, walking three metres, turning around, and then walking three metres back to chair and returning to the seated position. The TUG times will be noted down.

The extra measures besides the TUG test are questionnaires which will be given to patients to complete with the help of the Research Nurse.

The DEMQOL will involve carers completing the Carer part of the DEMQOL questionnaire. For those patients coming from nursing home's the nursing home staff will complete the DEMQOL carer questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-95 years
* Fresh unstable (AO/OTA type A2) pertrochanteric fracture
* If medically fit, patient will undergo surgical fixation within 48 hours of admission. Otherwise, all patients to be recruited must undergo surgery within 7 days of admission
* Patient or patient's carer/personal or nominated consultee has provided informed consent/assent to participate in the study
* Patient is considered able to complete the study assessment and visit schedule in the opinion of the investigating team

Exclusion Criteria:

* Unable to ambulate pre-injury, even with walking aids
* Unable to undergo surgical fixation within 7 days of admission
* Patient is for any reason considered unable to carry out the required study assessments or complete the follow-up visit schedule, in the opinion of the investigating team
* Previous stroke (non-recovered)
* Recent myocardial infarction (up to 60 days)
* Presence of fracture(s) in contralateral leg
* Presence of fracture(s) in ipsilateral leg, in addition to the pertrochanteric hip fracture
* Known renal or hepatic failure as defined by:

  * Elevated transaminases ≥ 2.0 x upper limits of normal for:

    * Serum aspartate aminotransferase (AST)
    * Serum alanine aminotransferase (ALT)
  * Significantly impaired renal function as determined by a derived creatinine clearance of ≤ 30 mL/min using the Modification of Diet in Renal Disease equation21

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
All patients attending week 4 follow-up visit must be able to perform the TUG test at least once. | 4 weeks
  The TUG test involves standing up from a seated position, walking three metres, turning around, and then walking three metres back to chair and returning to the seated position. The TUG times will be noted down in seconds/ minutes.

SECONDARY OUTCOMES:
The length of hospital stay for each patient | Average of 20 days
  Measure against the average of 20 days hospital stay after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giannoudis, MBBS,CCST,MD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No